CLINICAL TRIAL: NCT01802138
Title: A Pilot Study of Activated T Cell Therapy for Refractory/Relapsed Neuroblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILC_IIT_03
Record Dates: First submitted 2013-02-21; First posted 2013-03-01 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Neuroblastoma
Keywords: refractory/relapsed neuroblastoma patients
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Activated T-lymphocyte (Experimental): This was designed as a single-center, single group clinical trial, and subjects include patients with refractory refractory/relapsed neuroblastoma.
  If subjects agree to participate in the clinical trial by signing a written consent, only appropriate subjects, who meet the criteria on the examinations and tests, will undergo this clinical trial. To participate in the clinical trial, subject's blood of more than 60 ml should be withdrawn to make a study drug at least 3 weeks before administration. Subjects should visit to hospital according to the protocol and receive a study drug. Therapeutic response rate, overall survival rate, time to progression should be investigated.
  Interventions: Biological: Activated T lymphocyte

INTERVENTIONS:
Biological: Activated T lymphocyte — intravenous dripping of 200 ml (10^9~2*10^10 lymphocytes) for 1 hour.
  Other Names: Immuncell-LC

SUMMARY:
Activated T cell were manufactured through in vitro T cell expansion of autologous T cell. We designed this study to determine the feasibility and safety of Activated T-lymphocyte cell therapy for refractory/relapsed neuroblastoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 21 years or younger
* Histologically confirmed neuroblastoma
* Progressive disease after standard treatment or relapsed patient
* ECOG scale (ECOG-PS) ≤2
* Expected survival at least 3 months

Exclusion Criteria:

* Patients with autoimmune disease
* Patients with immunodeficiency
* Other malignancy 5 year prior to this study
* Severe organ dysfunction
* Severe allergic disease
* Severe psychiatric disorder
* Pregnancy or lactating woman

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
T cell count after in vitro expansion | up to 13 weeks
  T cell count after in vitro expansion
  Evaluation of safety

SECONDARY OUTCOMES:
Number of participants who showed response with Response Evaluation Criteria in Solid Tumors criteria | up to 1 year
  To determine the response rate
  To evaluate 1 yr progression free survival and overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea